CLINICAL TRIAL: NCT04902339
Title: Near-infrared Spectroscopy-based Neurofeedback as Adjunct to Mindfulness-Oriented Recovery Enhancement in Persons With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00129302
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain Syndrome; Opioid Use
MeSH Terms: interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MORE+NF (Experimental)
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement; Other: Neurofeedback
- MORE (Active Comparator)
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement
- Supportive Psychotherapy (Active Comparator)
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement — 8 weeks of therapy integrating mindfulness, reappraisal, and savoring skills.
  Arms: MORE; MORE+NF
Other: Neurofeedback — Near-infrared spectroscopy neurofeedback during savoring practice.
  Arms: MORE+NF
Behavioral: Supportive Psychotherapy — 8 weeks of supportive, process-oriented psychotherapy.
  Arms: Supportive Psychotherapy

SUMMARY:
The primary aim of this pilot trial is to enhance the efficacy of the Mindfulness-Oriented Recovery Enhancement (MORE) intervention by adding neurofeedback (NF) of the Orbitofrontal Cortex (OFC) as an adjunct to the savoring component of MORE. We hypothesize that the use of NF to train OFC responses during savoring will amplify patients' ability to savor and thereby increase brain responsivity to natural rewards; such enhanced reward responding will in turn be associated with improvements in clinical outcomes (e.g., pain, analgesic use).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age,
2. ability to understand and speak the English language
3. current chronic pain-related diagnosis

Exclusion Criteria:

1. mindfulness training experience (e.g., participation in MBSR/MBRP)
2. neurofeedback experience
3. current cancer diagnosis
4. having a psychiatric or medical condition that precludes the ability to provide informed consent or participation in outpatient treatment (e.g., psychosis, mania, acute intoxication)
5. suicidal ideation with a plan in the past week, or a suicide attempt in the past 3 months
6. unwilling, unable, or unlikely to complete study procedures (e.g., planned major surgery, anticipated move, travel barrier)
7. communication or cognitive impairment that limits participation in group treatment or study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) signaling | From baseline to immediately after the intervention.
  Changes in blood oxygenation levels to reward cues will be assessed, and planned comparisons will be performed between subjects receiving MORE+NF vs the control conditions.

SECONDARY OUTCOMES:
Opioid misuse | From baseline to 3-month follow-up.
  Scores on Current Opioid Misuse Measure, with higher scores indicating higher opioid misuse (min 0, max 68)
Chronic pain symptoms | From baseline to 3-month follow-up.
  Chronic pain symptoms will be measured with the Brief Pain Inventory, where higher scores indicate worse pain (min 0, max 10).
Opioid dose | From baseline to 3-month follow-up.
  Opioid dose as assessed with Timeline Followback Procedure
Savoring | From baseline to 3-month follow-up.
  Savoring as measured by the Brief Savoring Inventory, with higher scores indicating higher savoring (min 4, max 20)
Distress | From baseline to 3-month follow-up.
  Emotional distress measured by the Depression Anxiety Stress Scale-21, with higher scores indicating higher distress (min 0, max 63)
Self-transcendence | From baseline to 3-month follow-up.
  Self-transcendence measured by Nondual Awareness Dimensional Assessment, with higher scores indicating higher self-transcendence (min 13, max 65)
Pleasant sensation ratio | From baseline to immediately after intervention.
  Pleasant sensation ratio as measured by Sensation Manikin, a measure comprised of a visual body map to demonstrate the location and distribution of sensations.
Opioid craving | From baseline to 1-month follow-up.
  Opioid craving measured by numeric rating scale, with higher scores indicating worse craving (min 0, max 10)
Positive affect | From baseline to 1-month follow-up.
  Positive affect measured by numeric rating scale, with higher scores indicating higher positive affect (min 0, max 10)
Pleasure ratings | From baseline to immediately after intervention.
  Positive affect measured by numeric rating scale, with higher scores indicating higher pleasure (min 0, max 10)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garland, Principal Investigator — University of Utah
Locations (1):
- Center on Mindfulness and Integrative Health Intervention Development, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No